CLINICAL TRIAL: NCT07359417
Title: Improving Outcome of Patients With Squamous Cell ESophageal CArcinoma by Dose escaLATion Using High-prEcision Mr-guided Radiotherapy (ESCALATE): a Phase 1 Dose Finding Trial
Brief Title: MR-Guided Radiotherapy Dose Escalation Trial for Esophageal Squamous Cell Carcinoma
Acronym: ESCALATE
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: UMC Utrecht (Other)
Responsible Party: Principal Investigator, Stella Mook, Principal Investigator, UMC Utrecht
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NL86456.041.24
Record Dates: First submitted 2025-12-31; First posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2025-12

CONDITIONS: Esophageal Squamous Cell Carcinoma (ESCC); Esophageal Cancer, Squamous Cell
Keywords: MR-Guided Radiotherapy; Adaptive Radiotherapy; MR-Linac; Dose Escalation; Phase 1 Trial
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma

STUDY DESIGN:
Intervention Model Description: This is a phase 1 single-arm dose-escalation study using a 6+3 design with sequential patient cohorts treated at increasing radiotherapy dose levels.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental: MRI guided radiotherapy (Experimental): 2 sequential, homogenous boost fractions of 4-7 Gy on the gross tumor volume (GTV) in the week following CROSS using MR-guided online adaptive radiotherapy on the MRlinac.
  Start in dose level 0, of 2 x 5Gy boost per patient, and if safe this is increased step-wise to a maximum dose level 2 of 2 x 7Gy per patient.
  Interventions: Other: Radiation: MRI guided radiotherapy

INTERVENTIONS:
Other: Radiation: MRI guided radiotherapy — MRI guided radiotherapy
  Other Names: MRgRT; MR Linac

SUMMARY:
SUMMARY Rationale: Esophageal cancer (EC) is the seventh most frequently diagnosed cancer and the sixth leading cause of cancer-related death worldwide. As a result of the late onset of symptoms, most patients with EC present in an advanced stage with a corresponding poor prognosis. Poor disease outcome after surgery alone (5-yr overall survival between 25-40%) prompted many researchers to explore neoadjuvant chemoradiotherapy (nCRT) or neoadjuvant or perioperative chemotherapy (nCT/pCT) approaches. nCRT has led to pathological complete response (pCR) rate in squamous cell EC of almost 50%. Patients with a pCR have a favorable prognosis with 5-year OS >50%. In addition, patients who will achieve a pCR might be candidates for an organ preserving treatment strategy. Current standard nCRT consists of a relatively low dose of radiation compared to other tumors in the same area. The investigators hypothesize that increasing the dose of radiation will lead to increased local tumor control and pCR rates.

Objective: The main objective of this study is to determine the maximum tolerated dose (MTD) of 2-fraction boost MRI-guided radiotherapy (MRgRT) for patients with SCC following CROSS therapy. The secondary objectives are feasibility, non-dose limiting toxicity, oncological outcomes and to explore variables for early response evaluation.

Study design: 6+3 dose-escalation design with 3 radiotherapy dose levels. Study population: Patients with a resectable squamous cell esophageal carcinoma who are eligible for nCRT, surgery and MRgRT.

Intervention: 2 sequential, homogenous boost fractions of 4-7 Gy on the gross tumor volume (GTV) in the week following CROSS using MR-guided online adaptive radiotherapy on the MR-linac. Start in dose level 0, of 2 x 5Gy boost per patient, and if safe this is increased step-wise to a maximum dose level 2 of 2 x 7Gy per patient.

Main study parameters/endpoints: The primary endpoint is the incidence of a dose limiting toxicity (DLT). Early DLT is defined as radiation induced esophageal fistula/ perforation/ hemorrhage/ necrosis or tracheal, bronchial or bronchopleural fistula/tracheal or bronchopulmonary hemorrhage grade ≥ 3 or any non-hematological grade 4 toxicity according to Common Toxicity Criteria for Adverse Events (CTCAE) version 5.0 occurring within 14 weeks after the start of radiotherapy and before surgery or the postponing of surgery > 14 weeks after the end of radiotherapy due to any grade of treatment-related toxicity. Subacute DLT is defined as peri- and/or postoperative complications occurring within 30 days after surgery, defined as postoperative anastomotic leakage or pneumonitis ≥ 3b according to Clavien-Dindo. Secondary endpoints are non-DLT toxicity, the technical feasibility of dose delivery, perioperative complications, and oncological outcomes including R0 resection rate, histopathological tumor response, local and regional recurrence and death from any cause.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: The benefits for the patients may include higher probability of complete pathological response that initially leads to increased survival and could eventually result in organ-sparing treatment programs. Compared to standard treatment, the CROSS regimen including the sequential boost will take 2 days extra in the final week of CROSS. Possible risks include higher radiation toxicity and surgical complication rates. However, it is expected this increase to be minor, for the investigators will use dose constraints on organs at risk, which are associated with low radiation-induced toxicity, and they will not be exceeded.

ELIGIBILITY:
Inclusion criteria

In order to be eligible for this study, a subject must meet all of the following criteria:

* Histologically confirmed squamous cell carcinoma of the esophagus or GE- junction (Siewert I/II)
* Potentially resectable, locally advanced esophageal tumor (cT1bN+, cT2-3, N0-3, M0) based on standard primary staging by EUS and 18F-FDG PET-CT
* Scheduled to receive neoadjuvant chemoradiotherapy according to CROSS-regimen: weekly administration of carboplatin and paclitaxel for 5 weeks and concurrent radiotherapy (41.4Gy in 23 fractions, 5 days per week), followed by esophagectomy (as judged by the multidisciplinary tumor board)
* Tumor length ≤ 10 cm
* Age ≥ 18 years
* WHO performance status 0-2
* Signed informed consent
* Tumor volume that can be defined on MRI at baseline (T2w and DW-MRI)
* Absence of any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule before patient registration/randomization, written informed consent must be given according to ICH/GCP, and national/local regulations.

Exclusion criteria

A subject who meets any of the following criteria will be excluded from participation in this study:

* Adenocarcinoma of the esophagus
* Non-resectable, inoperable or metastatic squamous cell carcinoma of the esophagus or GE-junction
* Siewert type III
* Squamous cell carcinoma of the cervical esophagus
* Prior (chemo)radiotherapy to the mediastinum
* Prior esophageal surgery that impedes the ability to perform an esophagectomy
* Patients with multiple primary carcinomas of the esophagus
* Patients who meet exclusion criteria for MRI
* Irradical endoscopic mucosal resection (EMR) or endoscopic submucosal dissection (ESD) of primary tumor prior to start of neoadjuvant chemoradiotherapy
* Pregnant or breast-feeding patients
* Patients in whom it is not in their best interest to participate (in the judgment of the PI)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-05-30 (Actual); Primary Completion 2028-05-01 (Estimated); Study Completion 2028-05-01 (Estimated)

PRIMARY OUTCOMES:
Number of Participants Experiencing Dose-Limiting Toxicity (DLT) | From start of radiotherapy through 16 weeks after start of radiotherapy and up to 30 days after surgery
  Number of participants who experience a dose-limiting toxicity (DLT) after MR-guided radiotherapy, as defined in the study protocol. The maximum tolerated dose (MTD) will be determined as the highest radiotherapy dose level at which fewer than a predefined number of participants experience a DLT using a 6+3 dose-escalation design.

SECONDARY OUTCOMES:
Proportion of Participants Completing All Planned MR-Guided Radiotherapy Fractions | From start of radiotherapy through the end of the planned radiotherapy course (approximately 2 weeks)
  Feasibility of MR-guided radiotherapy, defined as the proportion of participants who complete all five planned radiotherapy fractions according to protocol without unplanned treatment discontinuation.
Pathological Tumor Response on Surgical Resection Specimen | At time of surgery
  Pathological response of the primary tumor and lymph node metastases assessed on the surgical resection specimen.
Disease-Free Survival | Up to 12 months after surgery
  Time from surgery to first documented disease recurrence or death from any cause.

CONTACTS AND LOCATIONS:
Locations (1):
- University Medical Center Utrecht, Utrecht, Utrecht, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided
Undecided. Plans for individual participant data (IPD) sharing have not been finalized at this time. Any future data sharing will depend on institutional policies, ethical approvals, and participant consent.